CLINICAL TRIAL: NCT02442076
Title: Skin and Acupuncture Needle Vibration Behaviors Through Observation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Central University,Taiwan(R.O.C) (Unknown)
Responsible Party: Principal Investigator, Chen Yu Sheng, Medical Doctor, Chang Gung Memorial Hospital
Other Study IDs: 103-5928A3
Record Dates: First submitted 2015-01-22; First posted 2015-05-13 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Skin Vibration; Acupuncture
Keywords: Skin vibration; Acupuncture needle vibration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Skin tremor induced by artery pulses are usually sensed by doctor's fingers in Traditional Chinese Medicine(TCM). On the other hand, vibration of acupuncture needle was also stated by Huang Di Nei Jing (Yellow Emperor). However; the characteristics of skin tremor and its correlation with vibrating acupuncture needles, how the skin tremor and vibration of needles varies from area to area, are not yet clarified.In this study, the abovementioned issues will be investigated experimentally through non-invasive method.

About 10 healthy volunteers, aged 20~65, will be recruited. The investigators will measure the needle and the skin tremor by video optical microscopy. The variation of skin tremor and needle vibration and their spectra will be analyzed digitally. The model correlating skin tremor, needle vibration and basic physiological parameters will be constructed.The fact that the skin tremor and the needle vibration come from the same origin is expected.

However; due to the leverage effects and different dynamical responses to the source vibrations at different frequencies, needle vibration might exhibit some difference from skin vibration in their power spectra. This study should be able to construct a clear model of the possible vibration sources such as heartbeat and breathing, the area dependence of vibrations, the correlation between the skin and the needle vibrations, and the correlation with other physiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy employees or students of National Central University aged between twenty to sixty-five.

Exclusion Criteria:

* With chronic diseases, severe psychological disorder or injury, or been in a surgery in the past twelve months.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers who is
  1. Aged 20~65
  2. Without chronic disease
  3. Didn't receive surgery in the past 12 months
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The frequency and spectra of the vibrating acupuncture needle ,by video optical microscopy | 30 minutes
The frequency and spectra of tremor of the skin surrounding the acupunctured point ,by video optical microscopy | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan